CLINICAL TRIAL: NCT03899792
Title: A Phase 1/2 Study of the Oral RET Inhibitor LOXO 292 in Pediatric Patients With Advanced RET-Altered Solid or Primary Central Nervous System Tumors
Brief Title: A Study of Oral LOXO-292 (Selpercatinib) in Pediatric Participants With Advanced Solid or Primary Central Nervous System (CNS) Tumors
Acronym: LIBRETTO-121
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17493; J2G-OX-JZJJ (Other: Eli Lilly and Company); LOXO-RET-18036 (Other: LOXO Oncology, Inc.); 2019-000212-28 (EudraCT Number)
Expanded Access: NCT03906331 (Approved for marketing)
Record Dates: First submitted 2019-02-06; First posted 2019-04-02 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Medullary Thyroid Cancer; Infantile Myofibromatosis; Infantile Fibrosarcoma; Papillary Thyroid Cancer; Soft Tissue Sarcoma
Keywords: Loxo; LOXO-292; KIF5B-RET; M918T; CCDC6-RET; RET-PTC1; NCOA4-RET; RET-PTC; RET-PTC3; RET-PTC4; PRKAR1A-RET; RET-PTC2; GOLGA5-RET; RET-PTC5; ERC1-RET; KTN1-RET; RET-PTC8; HOOK3-RET; PCM1-RET; TRIM24-RET; RET-PTC6; TRIM27-RET; TRIM33-RET; RET-PTC7; AKAP13-RET; FKBP15-RET; SPECC1L-RET; TBL1XR1-RET; BCR-RET; FGRF1OP-RET; RFG8-RET; RET-PTC9; ACBD5-RET; MYH13-RET; CUX1-RET; KIAA1468-RET; FRMD4A-RET; SQSTM1-RET; AFAP1L2-RET; PPFIBP2-RET; EML4-RET; PARD3-RET; G533C; C609F; C609G; C609R; C609S; C609Y; C611F; C611G; C611S; C611Y; C611W; C618F; C618R; C618S; C620F; C620R; C620S; C630R; C630Y; D631Y; C634F; C634G; C634R; C634S; C634W; C634Y; K666E; E768D; L790F; V804L; V804M; A883F; S891A; R912P; CLIP1-RET; Y806C; RET fusion; RET alteration; RET mutation; RET rearrangement; RET translocation; Neoplasms by Site; Neoplasms; Non-Small Cell Lung Cancer; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Cancer of Lung; Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Neoplasms, Pulmonary; Pulmonary Cancer; Pulmonary Neoplasms; Respiratory Tract Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Medullary Thyroid Cancer; Papillary Thyroid Cancer; Thyroid Diseases; Thyroid Neoplasms; Cancer of the Thyroid; Cancer of Thyroid; Neoplasms, Thyroid; Thyroid Adenoma; Thyroid Cancer; Thyroid Carcinoma; Endocrine System Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Thoracic Neoplasms; CNS tumor; Primary CNS tumor; Colonic Neoplasms; Cancer of Colon; Cancer of the Colon; Colon Cancer; Colon Neoplasms; Colonic Cancer; Neoplasms, Colonic; Malignant tumor of Breast; Mammary Cancer; Mammary Carcinoma, Human; Mammary Neoplasm, Human; Neoplasms, Breast; Tumors, Breast; Human Mammary Carcinoma; Malignant Neoplasm of Breast; Breast Carcinoma; Breast Tumors; Cancer of the Breast; Breast Neoplasms; Breast Cancer; RET Inhibitor; MTC; NSCLC; Soft tissue sarcoma; Infantile Myofibromatosis; Infantile Fibrosarcoma
MeSH Terms: conditions — Carcinoma, Medullary; Myofibromatosis; Thyroid Cancer, Papillary; Sarcoma; Neoplasms by Site; Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Tract Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Thyroid Diseases; Thyroid Neoplasms; Endocrine System Diseases; Endocrine Gland Neoplasms; Head and Neck Neoplasms; Thoracic Neoplasms; Central Nervous System Neoplasms; Colonic Neoplasms; Breast Neoplasms | interventions — selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Medullary Thyroid Cancer (MTC) Group (Experimental): Participants in this cohort had MTC and received 160 mg of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
  Interventions: Drug: Selpercatinib
- Cohort 2: Papillary Thyroid Cancer (PTC) Group (Experimental): Participants in this cohort had PTC and received 160 mg of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
  Interventions: Drug: Selpercatinib
- Cohort 3: Other Cancer Group (Experimental): Participants in this cohort had other (REarranged during Transfection (RET)-altered non-thyroid) cancer and received 160 mg of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
  Interventions: Drug: Selpercatinib

INTERVENTIONS:
Drug: Selpercatinib — Oral LOXO-292
  Other Names: LOXO-292; LY3527723

SUMMARY:
This is an open-label, multi-center Phase 1/2 study of oral LOXO-292 in pediatric participants with an activating rearranged during transfection (RET) alteration and an advanced solid or primary CNS tumor.

DETAILED DESCRIPTION:
This study includes 2 parts: phase 1 (dose escalation) and phase 2 (dose expansion). In phase 1, participants will be enrolled using a rolling 6 dose escalation scheme. The starting dose of LOXO-292 is equivalent to the adult recommended phase 2 dose of 160 milligrams (mg) twice a day (BID). Once the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) is identified, participants will be enrolled to one of four phase 2 dose expansion cohorts depending on tumor histology and tumor genotype. Cycle length will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid or primary CNS tumor which has failed standard of care therapies
* Evidence of an activating RET gene alteration in the tumor and/or blood
* Measurable or non-measurable disease
* Karnofsky (participants 16 years and older) or Lansky (participants younger than 16) performance score of at least 50
* Participant with primary CNS tumors or cerebral metastases must be neurologically stable for 7 days prior and must not have required increasing doses of steroids within the last 7 days
* Adequate hematologic, hepatic and renal function.
* Ability to receive study drug therapy orally or via gastric access
* Willingness of men and women of reproductive potential to observe conventional and effective birth control

Exclusion Criteria:

* Major surgery within two weeks prior to planned start of LOXO-292
* Clinically significant, uncontrolled cardiac, cardiovascular disease or history of myocardial infarction within 6 months prior to planned start of LOXO-292
* Active uncontrolled systemic bacterial, viral, fungal or parasitic infection
* Clinically significant active malabsorption syndrome
* Pregnancy or lactation
* Uncontrolled symptomatic hyperthyroidism or hypothyroidism (i.e. the participant required a modification to current thyroid medication in the 7 days before start of LOXO-292)
* Uncontrolled symptomatic hypercalcemia or hypocalcemia
* Known hypersensitivity to any of the components of the investigational agent, LOXO-292 or Ora-Sweet® SF and OraPlus®, for participants who will receive LOXO-292 suspension
* Prior treatment with a selective RET inhibitor(s) (including investigational selective RET inhibitor[s])

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2029-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (12):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - The Children's Hospital for Cancer and Blood Disorders, Aurora, Colorado
  - Nemours Children's Health, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Childrens Hospital, Houston, Texas
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Melbourne, Victoria
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Rigshospitalet, Copenhagen, Denmark
- Gustave Roussy, Villejuif, France
- Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Japan (4):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Kyoto University Hospital, Kyoto
- Seoul National University Hospital, Seoul, Korea, South Korea
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona], Spain
- University College Hospital - London, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of two parts: Phase 1 (dose-escalation) and Phase 2 (dose-expansion). In Phase 1, three participants received selpercatinib, with dosing based on body surface area. The starting dose level was 92 mg/m^2 (maximum 160 mg, twice daily (BID]), selected to approximate the exposure associated with the recommended Phase 2 dose (RP2D) in adults. The Phase 2 portion opened for enrollment after confirmation of the RP2D of 92 mg/m^2 (maximum 160 mg BID).
Pre-assignment Details: In Phase 2, participants were assigned to one of three disease-based groups: medullary thyroid cancer (MTC), papillary thyroid cancer (PTC), or Other Solid Tumors and received selpercatinib at the RP2D. Current primary results are reported, and additional results will be reported during study completion.
Groups:
- Dose Escalation Cohort (Phase 1): Participants received selpercatinib given orally BID, with the dose based on body surface area in a 28-day cycle. The starting dose level of 92mg/m^2 BID (maximum160 mg BID) was intended to deliver equivalent exposure to the RP2D in adults.
- Cohort 1 (Phase 2): Medullary Thyroid Cancer (MTC) Group: Participants in this cohort had MTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Cohort 2 (Phase 2): Papillary Thyroid Cancer (PTC) Group: Participants in this cohort had PTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Cohort 3 (Phase 2): Other Cancer Group: Participants in this cohort had other (RET-altered non-thyroid) cancer and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
Period: Phase 1
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1 (Phase 2): Medullary Thyroid Cancer (MTC) Group | Cohort 2 (Phase 2): Papillary Thyroid Cancer (PTC) Group | Cohort 3 (Phase 2): Other Cancer Group
Started | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1 (Phase 2): Medullary Thyroid Cancer (MTC) Group | Cohort 2 (Phase 2): Papillary Thyroid Cancer (PTC) Group | Cohort 3 (Phase 2): Other Cancer Group
Started | 0 | 15 (Out of 15 participants, 2 participants transitioned from Phase 1.) | 15 | 6 (Out of 6 participants, 1 participant transitioned from Phase 1.)
Received At Least 1 Dose of Study Drug | 0 | 15 | 15 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 15 | 15 | 6
Not completed — Ongoing Treatment | 0 | 13 | 14 | 2
Not completed — Death | 0 | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug. The Baseline data were planned to be presented according to Phases. Here "number analyzed" signifies participants who were evaluable for specified Phase of the study.
Groups:
- Dose Escalation Cohort (Phase 1): Participants received selpercatinib given orally BID, with the dose based on body surface area in a 28-day cycle. The starting dose level of 92mg/m^2 (maximum160 mg BID) was intended to deliver equivalent exposure to the RP2D in adults.
- Cohort 1 (Phase 2): MTC Group: Participants in this cohort had MTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Cohort 2 (Phase 2): PTC Group: Participants in this cohort had PTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Cohort (Phase 1) | Cohort 1 (Phase 2): MTC Group | Cohort 2 (Phase 2): PTC Group | Cohort 3 (Phase 2): Other Cancer Group | Total
Number analyzed (Participants) | 3 | 13 | 15 | 5 | 36
Age, Customized [Count of Participants; unit: Participants]
  Age: <=18 years | 2 | 10 | 13 | 5 | 30
  Age: Between 18 and 65 years | 1 | 3 | 2 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented according to Phases. Here "number analyzed" signifies participants who were evaluable for specified Phase of the study.
  Participants
    Female | 2 | 5 | 7 | 3 | 17
    Male | 1 | 8 | 8 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented according to Phases. Here "number analyzed" signifies participants who were evaluable for specified Phase of the study.
  Participants
    Hispanic or Latino | 3 | 0 | 4 | 0 | 7
    Not Hispanic or Latino | 0 | 11 | 11 | 4 | 26
    Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Baseline data were planned to be presented according to Phases. Here "number analyzed" signifies participants who were evaluable for specified Phase of the study.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 7 | 3 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 2 | 0 | 0 | 2
    White | 3 | 9 | 6 | 0 | 18
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 2 | 2 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 2 | 2 | 1 | 5
  South Korea | 0 | 0 | 4 | 2 | 6
  United States | 3 | 3 | 4 | 1 | 11
  Japan | 0 | 0 | 2 | 1 | 3
  Denmark | 0 | 1 | 0 | 0 | 1
  Italy | 0 | 0 | 2 | 0 | 2
  France | 0 | 1 | 0 | 0 | 1
  Australia | 0 | 4 | 0 | 0 | 4
  Germany | 0 | 2 | 0 | 0 | 2
  Spain | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was any of the adverse events that starts on or after the first administration of study drug listed below, as defined by the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
  * Any Grade(G) ≥3 nonhematologic toxicity except G3 fatigue, nausea, tendon reflex decrease, weight gain attributable to normal growth and development.
  * G3 vomiting/diarrhea was DLT only if it persists >48 h despite standard of care treatment.
  * G4 vomiting/diarrhea was DLT regardless of duration.
  * Any toxicity, regardless of the NCI CTCAE v5.0 grade, resulting in discontinuation or dose reduction of treatment (except symptoms related to progressive disease (PD)).
  * G4/G3 thrombocytopenia with G1 or higher bleeding.
  * G4 anemia lasting >8 days, despite supportive therapy.
  * G4 neutropenia, lasting >8 days, despite supportive therapy
Time Frame: Cycle 1 (28 Day Cycle)
Population: All participants in Phase 1 of the study who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Cohort (Phase 1)
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Phase 2: Percentage of Participants With Overall Response Rate (ORR) in Study
Description: ORR: Percentage of participants who achieve best overall response Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST).
  * CR is defined as disappearance of all target lesions.
  * PR is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: Date of first dose to disease progression or death (Up to 62.4 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (Phase 2): MTC Group | Cohort 2 (Phase 2): PTC Group | Cohort 3 (Phase 2): Other Cancer Group
Number analyzed (Participants) | 15 | 15 | 6
Percentage of participants | 60.0 | 53.3 | 33.3

3. Secondary Outcome: Plasma Concentrations of LOXO-292
Description: Outcome data will be provided after the study is completed.
Time Frame: Days 1 and 8 of Cycle 1, Day 1 of Cycle 3 and Day 8 after Intra-participant Dose Escalation (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2029-05

4. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 24 Hours (AUC0-24) of LOXO-292
Description: Outcome data will be provided after the study is completed.
Time Frame: Days 1 and 8 of Cycle 1, Day 1 of Cycle 3 and Day 8 after Intra-participant Dose Escalation (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2029-05

5. Secondary Outcome: Maximum Concentration (Cmax) of LOXO-292
Description: Outcome data will be provided after the study is completed.
Time Frame: Days 1 and 8 of Cycle 1, Day 1 of Cycle 3 and Day 8 after Intra-participant Dose Escalation (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2029-05

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of LOXO-292
Description: Outcome data will be provided after the study is completed.
Time Frame: Days 1 and 8 of Cycle 1, Day 1 of Cycle 3 and Day 8 after Intra-participant Dose Escalation (each cycle is 28 days)
Reporting Status: Not Posted, anticipated posting 2029-05

7. Secondary Outcome: Recommended LOXO-292 Dose for Phase 2 (MTD)
Description: Outcome data will be provided after the study is completed.
Time Frame: Cycle 1 (28 days)
Reporting Status: Not Posted, anticipated posting 2029-05

8. Secondary Outcome: To Assess the Preliminary Anti-Tumor Activity of LOXO-292 in Pediatric Participants With Tumors Harboring an Activating RET Alteration as Determined by ORR Based on RECIST v1.1
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline to Progressive Disease or Death due to any cause (Estimated up to 12 months)
Reporting Status: Not Posted, anticipated posting 2029-05

9. Secondary Outcome: Changes From Baseline in Pain Measures as Measured by Wong Baker Faces Scales. Wong-Baker Faces Pain Scale Includes Pictures of Facial Expressions With Correlating Scores of 0 Being 'no Hurt' and 10 Being 'Hurts Worst'.
Description: Outcome data will be provided after the study is completed.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2029-05

10. Secondary Outcome: Changes From Baseline in Health Related Quality of Life Measures as Measured by Pediatric Quality of Life (PedsQoL) Inventory Core. PedsQoL Includes a List of Problems With Scores of 0 Being 'Never a Problem' and 4 Being 'Almost Always a Problem'.
Description: Outcome data will be provided after the study is completed.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2029-05

11. Secondary Outcome: Objective Response Rate as Assessed by RECIST v1.1, as Assessed by Investigator
Description: Outcome data will be provided after the study is completed.
Time Frame: Approximately every 8 weeks for one year, then every 12 weeks, and 7 days after the last dose (for up to 2 years) in participants who have not progressed.
Reporting Status: Not Posted, anticipated posting 2029-05

12. Secondary Outcome: Objective Response Rate as Assessed by RANO, as Assessed by Investigator
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

13. Secondary Outcome: Duration of Response (DOR) as Assessed by Investigator
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

14. Secondary Outcome: Duration of Response (DOR) as Assessed by the IRC
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

15. Secondary Outcome: Progression Free Survival (PFS) as Assessed by Investigator
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

16. Secondary Outcome: PFS as Assessed by IRC
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

17. Secondary Outcome: Overall Survival (OS)
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 11
Reporting Status: Not Posted, anticipated posting 2029-05

18. Secondary Outcome: Clinical Benefit Rate (by Investigator)
Description: Outcome data will be provided after the study is completed.
Time Frame: Approximately every 8 weeks for one year, then every 12 weeks, 7 days after the last dose (for up to 2 years) in participants who have not progressed.
Reporting Status: Not Posted, anticipated posting 2029-05

19. Secondary Outcome: Clinical Benefit Rate (by IRC)
Description: Outcome data will be provided after the study is completed.
Time Frame: as for outcome 18
Reporting Status: Not Posted, anticipated posting 2029-05

20. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Outcome data will be provided after the study is completed.
Time Frame: From the time of informed consent, for approximately 24 months (or earlier if the participants discontinues from the study), and through Safety Follow-up (28 days after the last dose)
Reporting Status: Not Posted, anticipated posting 2029-05

21. Secondary Outcome: To Evaluate the Concordance of Prior Molecular That Detected a RET Alteration Within the Participant's Tumor With Diagnostic Tests Being Evaluated by Sponsor
Description: Outcome data will be provided after the study is completed.
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2029-05

22. Secondary Outcome: Phase 2: Post-Operative Stage on Participants Treated With LOXO-292
Description: Tumor stage is described according to the Tumor, Node, Metastasis (TNM)Classification of malignant tumors of the Union for International Cancer Control (UICC). Outcome data will be provided after the study is completed.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2029-05

23. Secondary Outcome: Phase 2: Surgical Margin Status in Participants Treated With LOXO-292
Description: Tumor margins after surgery are classified into four groups using the International Cancer Control (UICC)-R classification and the Intergroup Rhabdomyosarcoma Staging (IRS) systems: 1) Complete tumor resection with histologically free margins, 2) Macroscopic resection but invaded margins on histology, 3)Macroscopic residual tumor and 4) Distant metastatic tumor. Outcome data will be provided after the study is completed.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2029-05

24. Secondary Outcome: Descriptive Analysis of Pretreatment Surgical Plan
Description: Outcome data will be provided after the study is completed.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2029-05

25. Secondary Outcome: Descriptive Analysis of Post-Treatment Plans
Description: Outcome data will be provided after the study is completed.
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2029-05

ADVERSE EVENTS:
Time Frame: Baseline up to 64 months
Description: The Safety Analysis data presented for overall population irrespective of phases. All participants who received at least one dose of the study drug. Per prespecified analysis plan, all Phase 1 and Phase 2 participants were planned to be analyzed together for Adverse events and Mortality data.
Groups:
- Cohort 1: MTC Group: Participants in this cohort had MTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Cohort 2: PTC Group: Participants in this cohort had PTC and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
- Cohort 3: Other Cancer Group: Participants in this cohort had other (RET-altered non-thyroid) cancer and received 92mg/m^2 (maximum160 mg BID) of selpercatinib BID orally on Days 1 through 28 of a 28-day cycle.
  The treatment was continued until participants experienced a progressive disease, unacceptable toxicity, or other protocol-defined reason for discontinuation.
Arm/Group | Cohort 1: MTC Group | Cohort 2: PTC Group | Cohort 3: Other Cancer Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 4/6
Serious Adverse Events (participants affected / at risk) | 8/15 | 4/15 | 3/6
Other Adverse Events (participants affected / at risk) | 15/15 | 15/15 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MTC Group (N=15) | Cohort 2: PTC Group (N=15) | Cohort 3: Other Cancer Group (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: MTC Group (N=15) | Cohort 2: PTC Group (N=15) | Cohort 3: Other Cancer Group (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 (15) | 1 (1) | 2 (4)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 3 (4) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (2) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (11) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (4) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (12) | 2 (2) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (13) | 10 (26) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (12) | 5 (15) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 9 (18) | 2 (8) | 0 (0)
Asthenia (General disorders) | 1 (3) | 2 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Face oedema (General disorders) | 4 (4) | 1 (3) | 1 (1)
Fatigue (General disorders) | 4 (8) | 4 (8) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (4) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Medical device site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (4) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 7 (13) | 4 (4) | 3 (7)
Swelling (General disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Aeromonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 6 (8) | 4 (5) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (2) | 0 (0)
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Moraxella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (3) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pathogen resistance (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (5) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (16) | 2 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (5) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (6) | 5 (9) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 3 (7) | 8 (13) | 3 (4)
Blood 1,25-dihydroxycholecalciferol decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 2 (4) | 2 (2)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (26) | 3 (45) | 2 (3)
Blood calcitonin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (3) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (7) | 0 (0)
Blood creatinine increased (Investigations) | 2 (4) | 3 (7) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 4 (10) | 1 (1) | 2 (3)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 3 (5) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qrs complex prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 2 (6) | 1 (4) | 1 (1)
Electrocardiogram t wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Haemoglobin increased (Investigations) | 1 (3) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (4) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (5) | 0 (0) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (21) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pregnancy test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Thyroglobulin increased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Urine analysis abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin d decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight increased (Investigations) | 4 (9) | 3 (5) | 0 (0)
White blood cell count decreased (Investigations) | 3 (7) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2) | 1 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (15) | 3 (4) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (28) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (13) | 2 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (8) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (20) | 2 (2) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sever's disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 4 (8) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Nitrituria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 2 (4) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (4) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0)
Ovarian rupture (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (5) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 2 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (7) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (7) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dental operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (10) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2025-02-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03899792/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT03899792/SAP_001.pdf